CLINICAL TRIAL: NCT02603315
Title: To Assess the Correlation Between the Predictive Factor of Vascularity (CD74) in Malignant Pleural Mesothelioma and Treatment Results (Response Rate, and Overall Survival )
Brief Title: Vascularity Impact on the Treatment Outcome in Malignant Pleural Mesothelioma(VITMPM)
Acronym: VITMPM
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Muna Sami Jassim, Doctor in clinical oncology and nuclear medicine department, Ain Shams University
Other Study IDs: DR-81
Record Dates: First submitted 2015-10-28; First posted 2015-11-11 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2015-10

CONDITIONS: Malignant Pleural Mesotheliomas
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Vascular Endothelial Growth Factor A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: marker CD74 and vascular endothelial growth factor VEGF — correlate the result of vascularity test done on paraffin blocks on both types of malignant pleural mesothelioma patients diagnosed and receive treatment and evaluated after treatment

SUMMARY:
The purpose of this study is to To assess the correlation between the predictive factor of vascularity (CD74) in malignant pleural mesothelioma and treatment results (response rate, and overall survival) .

DETAILED DESCRIPTION:
This is a randomized controlled retrospective study through Examination of paraffin blocks of the patient selected to be included in the study for assessment of the selected vascularity marker of malignant pleural mesothelioma of both types . The CD74 (LN2) antibody is intended for qualified laboratories to qualitatively identify by light microscopy the presence of associated antigens in sections of formalin-fixed paraffin-embedded tissue sections using Immunohistochemistry test methods.

ELIGIBILITY:
Inclusion Criteria:

* Histopathological confirmation of malignant pleural mesothelioma .
* Full clinical data.
* Availability for follow up: Personal communication will be attempted in order to collect missing information.

  3-The files of all patients will be reviewed to analyze the following :
* Operative data if done .
* Pathological review and immunohistochemistry.
* Laboratory investigations: (routine investigations: complete blood picture,liver and renal function test)
* Radiological investigations:( CXR and CT-chest, Abdominal and pelvic U\S and MRI ).
* Treatment protocols applied: Radiotherapy and Chemotherapy.
* Response and survival after treatment .

Exclusion Criteria:

* cases not receive chemotherapy ,on available of evaluation after treatment

Ages: 39 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Egyptian patients with confirmed malignant pleural mesothelioma
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-10; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
to correlate the results of the vascularity marker of pleural mesothelioma CD74 of patients attended to Ain Shams University hospitals with the result response of treatment by chemotherapy ,overall survival and progreeion free survival | 3-4 months
  The cases diagnosed and receive at the least 2-3 cycles of chemotherapy and evaluated after treatment

SECONDARY OUTCOMES:
assessment of vascular enothelial growth factor (VEGF) in patient with malignant pleural mesothelioma who attended to Ain Shams University and made comparison with the result of CD 74 | 3-4 months
  The cases diagnosed and receive at the least 2-3 cycles of chemotherapy and evaluated after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Amr S Saad, MD, Study Director — Ain Shams University; Mahmoud Ellithy, MD, Study Chair — Ain Shams University; Doaa Atef, MD, Study Director — Ain Shams University; Hoda Abougabal, MD, Study Director — Ain Shams University
Locations (1):
- Ain Shams University Hospital, Cairo, Egypt